CLINICAL TRIAL: NCT07194538
Title: One-Year Follow-Up of Clinical and Tomographic Parameters After Conventional (3 mW/cm² × 30 Min) Versus Accelerated (9-10 mW/cm² × 10 Min) Epi-Off Corneal Collagen Cross-Linking
Brief Title: One-Year Outcomes After Conventional vs Accelerated Epi-Off Corneal Cross-Linking in Progressive Keratoconus (Observational Cohort)
Acronym: KCXL-1Y
Status: Completed | Type: Observational
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Iva Bešlić, Medical Doctor, Ophtalmology and Optometrist Specialist, FEBO, Clinical Hospital Centre Zagreb
Other Study IDs: 8.1-25/223-2 02/013 AG
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Keratoconus
Keywords: keratoconus; corneal crosslinking; conventional CXL; accelerated CXL; ABCD grading system; one-year outcome; Scheimpflug tomography
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 - CXL30 (Conventional): Conventional Dresden protocol; irradiance 3 mW/cm² for 30 minutes; epi-off; riboflavin 0.1%. Assignment was per treating surgeon's standard-of-care decision (no prospective allocation).
- Cohort 2 - CXL10 (Accelerated): Accelerated protocol; irradiance 9 mW/cm² for 10 minutes; epi-off; riboflavin 0.1%. Assignment was per treating surgeon's standard-of-care decision (no prospective allocation).

SUMMARY:
Prospective, observational (consecutive eligible eyes) continuation of a previously published 6-month cohort from the same center, extending follow-up to 12 months. Patients with progressive keratoconus received either conventional (CXL30: 3 mW/cm² × 30 min) or accelerated (CXL10: 9 mW/cm² × 10 min) epi-off CXL as part of routine clinical care. Assignment to CXL30 or CXL10 was at the discretion of the treating surgeon; no prospective allocation or randomization was performed. Outcomes included ABCD grading metrics (ABCD-A/B), Kmax, anterior/posterior radii of curvature (ARC/PRC), thinnest pachymetry, and visual acuity at 12 months. The primary objective was to evaluate one-year stabilization/remodeling and compare anterior/posterior responses between protocols.

DETAILED DESCRIPTION:
This prospective, single-center observational cohort extends the follow-up of a previously reported 6-month series from the same center to a 12-month horizon. The study population comprises consecutive patients with progressive keratoconus managed with standard-of-care, epi-off corneal collagen cross-linking (CXL) at the University Hospital Centre Zagreb. Patients were treated according to routine clinical decision-making by the attending surgeon; no prospective allocation or randomization to a protocol was performed. In routine care, some eyes underwent conventional CXL30 (Dresden-type; UVA 370 nm, 3 mW/cm² for 30 min) and others underwent CXL10 (accelerated; UVA 370 nm, 9 mW/cm² for 10 min). Riboflavin 0.1% solution was used per institutional practice. All procedures were epi-off.

Rationale. While both conventional and accelerated CXL are widely used in daily practice, comparative one-year data that integrate tomographic metrics from the ABCD grading system with traditional surrogates (e.g., Kmax) help clarify the balance between anterior corneal flattening, posterior remodeling, and pachymetric behavior under real-world conditions. This observational design captures effectiveness and safety without altering clinical decision pathways.

Design and cohorts. Consecutive eligible eyes were enrolled at the time of surgery and followed prospectively at baseline (day of surgery) and 1, 3, 6, and 12 months. Two observational cohorts are defined post hoc by the protocol actually received in standard care:

CXL30 (Conventional): continuous UVA 3 mW/cm² × 30 min (Dresden-type).

CXL10 (Accelerated): continuous UVA 9 mW/cm² × 10 min.

Assignment to CXL30 vs CXL10 was at the surgeon's discretion based on routine clinical considerations; the study did not prospectively assign interventions.

Eligibility. Inclusion required progressive keratoconus documented on serial Scheimpflug tomography within the prior 12 months; a clear corneal axis (no visually significant scarring); and corneal thickness 370 µm or more per institutional safety protocol. Exclusions comprised no central corneal scars, prior chemical burns, severe corneal infection, or ocular surface disease. Pregnancy and lactation during treatment were also contraindications.

Examinations and outcomes. Outcomes were assessed using Scheimpflug tomography (e.g., Pentacam or equivalent) and standard visual testing. The primary outcome was change in ABCD-A (anterior corneal curvature metric) from baseline to 12 months. Secondary outcomes included Kmax, anterior and posterior radii of curvature (ARC/PRC), thinnest pachymetry, and UDVA/BCVA at 12 months. Safety endpoints encompassed delayed epithelial healing (>7 days), infectious keratitis, clinically significant corneal haze, endothelial decompensation, and need for re-treatment.

Follow-up timeline. Enrollment/treatment occurred May 2021-December 2021; 12-month follow-up was completed by January 2023. Of the 28 eyes in the previously reported 6-month cohort, 22 completed the 12-month visit and were included in this analysis.

Data handling and oversight. Data were collected prospectively in a standardized fashion and analyzed as observational (no masking, no allocation). The protocol was reviewed and approved by the institutional Ethics Committee; all analyses used de-identified data. No data monitoring committee was required given the non-interventional, standard-of-care nature of the study.

Statistical approach (summary). Effectiveness outcomes are summarized descriptively; within-cohort change from baseline to 12 months is evaluated with paired tests on continuous variables as appropriate to distributional assumptions. Between-cohort comparisons (CXL30 vs CXL10) at 12 months and for change scores are explored with two-sample tests or generalized linear models with adjustment for prespecified covariates (e.g., baseline severity indices) where applicable. Statistical significance is assessed at a two-sided α = 0.05, with corresponding confidence intervals to aid interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Progressive keratoconus documented on serial Scheimpflug tomography within the prior 12 months (ABCD/K-metrics and/or pachymetry).
* Clear corneal axis (no visually significant scarring).
* Corneal thickness 370 μm or more

Exclusion Criteria:

* No central corneal scars, prior chemical burns, severe corneal infection, or ocular surface disease.
* No pregnancy and lactation during treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with progressive keratoconus treated at University Hospital Centre Zagreb (Croatia).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-05-09 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Change in ABCD-A from baseline to 12 months | 12 months
  Belin ABCD parameter A = A stage (ordinal severity stage); Belin ABCD keratoconus grading system (A = anterior corneal radius of curvature at the thinnest point; B = posterior corneal radius of curvature at the thinnest point; C = thinnest corneal pachymetry; D = distance best-corrected visual acuity).
  minimum value 0, maximum value 4 (ordinal scale 0-4) higher score means worse outcome

SECONDARY OUTCOMES:
Change in ARC from baseline to 12 months | 12 months
  ABCD A = ARC; mm ARC - anterior radius curvature calculated from a 3.0 mm optical zone centered on the thinnest point of the cornea higher = flatter (better); mm
Change in PRC from baseline to 12 months | 12 months
  PRC; mm PRC - posterior radius curvature calculated from a 3.0 mm optical zone centered on the thinnest point of the cornea higher = flatter (better); mm Time Frame: 12 months
Change in Kmax from baseline to 12 months | 12 months
Change in UDVA and BCVA from baseline to 12 months | 12 months
  UDVA = uncorrected visual acuity ; BVCA = best corrected visual acuity
Change in thinnest pachymetry from baseline to 12 months | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Centre Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No
Individual participant datasets will not be shared. The informed consent and IRB approval did not include permission for public sharing of participant-level data, and the small, single-center cohort with imaging-derived variables carries a residual re-identification risk. De-identified aggregate results and summary tables will be available in the published article and can be provided upon reasonable request to the corresponding author, subject to institutional approvals.